CLINICAL TRIAL: NCT05794724
Title: Concordance Between Intraoperative Frozen Section Pathology and Postoperative Paraffin-embedded Pathology in Diagnosing Spread Through Air Space (STAS) of Lung Adenocarcinoma
Brief Title: Intraoperative Frozen Section Pathology to Guide Surgical Treatment for Lung Adenocarcinoma (ECTOP-1016)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Other Study IDs: CONCORD-C
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Lung Adenocarcinoma; Surgical Procedure, Unspecified; Pathology
Keywords: Intraoperative frozen section pathology; Surgical treatment; Lung adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical T1N0M0 lung adenocarcinoma patients eligible for surgery.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection of lung adenocarcinoma. Wedge resection, segmentectomy or lobectomy will be performed according to each patients' condition.

SUMMARY:
This study is one of Eastern Cooperative Thoracic Oncology Projects (ECTOP-1016). The goal of this clinical trial is to confirm the concordance rate between intra-operative frozen section pathological diagnosis and post-operative paraffin embedded pathological diagnosis, and use this result to guide surgical treatment for early stage (cT1N0M0) lung adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent form and are willing to complete the study according to the study protocol;
* No previous history of cancer or pulmonary surgery;
* Solitary lesions or multiple lesions with only one not manifesting as pure ground-glass opacity (GGO) on CT scan;
* Peripheral clinical T1N0M0 patients that are eligible for surgery;
* Non-small cell lung cancer is pathologically diagnosed before or at surgery;
* No radiation therapy or chemotherapy before surgery.

Exclusion Criteria:

* Patients with clinical stages other than T1N0M0;
* The lesion cannot be completely resected;
* Previous history of cancer;
* Patients having received radiation therapy or chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical stage T1N0M0 lung adenocarcinoma patients who are going to undergo surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of spread through air space (STAS).

SECONDARY OUTCOMES:
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of IASLC grades of lung adenocarcinoma
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of lung adenocarcinoma subtypes according to the WHO classifications.
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of pleural invasion and lymph node invasion.
Recurrence-free survival (RFS) | 5 years
  Recurrence-free survival (RFS)
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the time from date of curative surgery to the time of death of any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided